CLINICAL TRIAL: NCT05746182
Title: Genetic Predisposition Testing Program for Pancreatic Neuroendocrine Neoplasms
Acronym: PanNEN
Status: Recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: University of California Pancreatic Cancer Consortium (UCPCC) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 224513; NCI-2023-01566 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2023-02-17; First posted 2023-02-27 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Neuroendocrine Neoplasm
Keywords: Genetic Assay; Biomarkers
MeSH Terms: conditions — Adenoma, Islet Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva samples will be obtained from participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with Pancreatic Neuroendocrine Neoplasms
  Interventions: Diagnostic Test: Hereditary Cancer Panel

INTERVENTIONS:
Diagnostic Test: Hereditary Cancer Panel — UCSF's Internal Clinical Laboratory Improvement Amendments of 1988 (CLIA)-certified Expanded Hereditary Cancer Panel will be employed which measures a minimum 88 genes
  Other Names: University of California, San Francisco's (UCSF) Expanded Hereditary Cancer Panel; Germline Testing

SUMMARY:
This is a prospective observational multi-center pilot study of germline testing for participants receiving care at University of California participating locations with a new or existing diagnosis of Pancreatic Neuroendocrine Neoplasms (PanNEN). This protocol is an extension of existing Genetic Testing Station efforts at University of California, San Francisco (UCSF)

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the frequency of germline mutations in patients with PanNEN.

SECONDARY OBJECTIVES:

I. To assess the rates of different types of germline mutations in patients PanNEN.

II. To assess the rates of different types of variants of uncertain significance in patients with PanNEN.

III. To estimate the rate of completion of genetic testing in patients who are offered prospective germline testing.

EXPLORATORY OBJECTIVES:

I. To examine attitudes of patients who have completed germline testing.

II. To explore reasons for declining germline testing.

III. In patients with repeat germline testing, compare the frequency of germline alteration between tests.

IV. Assess the relationship between germline pathogenic variants and somatic mutations in PanNEN.

OUTLINE:

Potential eligible participants will be identified via chart review and invited to consent to the study. Study participants who agree to prospective testing and have not had previous large panel germline testing will watch an informational video about germline testing and be offered testing with University of California, San Francisco's (UCSF) Expanded Hereditary Cancer Panel. Study participants who decline germline testing will be asked to answer a one-question Declination Survey. Results will be shared with participants and their providers per the standard of practice at each participating study site. All participants who decided to receive germline testing will be asked to complete a decision survey.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed PanNEN.

   a. The diagnostic biopsy may have been taken from any site (primary or metastatic).
2. New and existing PanNEN participants will be eligible (any grade, any stage, any age > 18 years).
3. Participants willing and able to comply with the study procedures.

Exclusion Criteria:

1. Inability to provide informed consent.
2. For participants who have not had prior testing with a dedicated germline pane of at least 80 genes:

   1. Inability to speak/read a language supported by the germline testing station (GTS). The supported languages currently include English, Korean, Japanese, Vietnamese, Russian, Tagalog, Farsi, Spanish, Cantonese, Mandarin, and Arabic).
   2. Active hematologic malignancy.
   3. History of allogenic bone marrow transplant or stem cell transplant.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All participants receiving care at University of California participating locations with a new or existing diagnosis of PanNEN
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-04-07 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of overall pathogenic germline mutations | Up to 2 years
  The overall percentage of participants with pathogenic, or likely pathogenic germline mutations will be reported with 95% confidence intervals

SECONDARY OUTCOMES:
Rates of different types of pathogenic mutations | Up to 2 years
  The percentage of participants with each identified type of pathogenic, or likely pathogenic, will be reported with 95% confidence intervals
Rates of different types of variants of uncertain significance (VUS) | Up to 2 years
  The percentage of participants with identified variants of uncertain significance will be reported with 95% confidence intervals.
Rate of declination for participants offered testing. | Up to 2 years
  Participants who decline genetic testing but agree to participate in other study procedures will complete a Declination Survey which consists of one questions asking the reason for the decision to decline germline testing.
Rate of completion of testing | Up to 2 years
  The rate of study completion defined as the percentage of participants who agree to testing, and complete all study procedures through return of results and meeting with genetic counselor (as appropriate) will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Bergsland, MD, Principal Investigator — University of California, San Francisco
Locations (3):
- United States (3):
  - University of California, Los Angeles, Los Angeles, California
  - Univeristy of California, San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: No